CLINICAL TRIAL: NCT03908814
Title: Phase I Clinical Trial to Evaluate the Safety, Tolerance and Pharmacokinetics of Human Anti-PD-L1 Monoclonal Antibody Injection (LDP) in Patients With Advanced Malignant Tumors
Brief Title: Phase I Clinical Trial of Human Anti-PD-L1 Antibody Injection (LDP) in Patients With Advanced Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dragonboat Biopharmaceutical Company Limited (Industry)
Collaborators: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LDP100001
Record Dates: First submitted 2019-04-08; First posted 2019-04-09 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-04

CONDITIONS: Advanced Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug: LDP (Experimental): This is a dose-escalation trial, all participants will receive treatment with LDP. Participants enrolled in this trial may receive one of the following doses dependent upon time of enrolment into the study.
  Cohort 1: 0.1 mg/kg Cohort 2: 0.3 mg/kg Cohort 3: 1 mg/kg Cohort 4: 3 mg/kg Cohort 5: 10 mg/kg Cohort 6: 10 mg/kg
  Interventions: Drug: Whole Human Anti-PD-L1 Antibody Injection (LDP)

INTERVENTIONS:
Drug: Whole Human Anti-PD-L1 Antibody Injection (LDP) — Dose escalation study evaluating six dose levels (0.1, 0.3, 1, 3 , 10and 20 mg/kg) of LDP.
  Other Names: LDP

SUMMARY:
This is a phase I, open-label, multiple-dose, dose-escalation study to evaluate the safety, tolerability, pharmacokinetics and anti-tumor activity of LDP in subjects with advanced malignant tumors.

DETAILED DESCRIPTION:
This trial is an open, dose escalation phase I clinical trial study of patients with advanced cancer who have failed standard treatment. The trial is divided into a dose escalation phase and an expansion phase.

Approximately 130 patients will be enrolled in this trial. The dose-increasing phase is about 30 cases, and the expansion stage is about 100 cases.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 (inclusive), regardless of gender
2. Histologically or cytologically confirmed patients with advanced malignant tumors who fail to receive standard treatment or have no standard treatment or are not suitable for standard treatment at this stage;
3. The estimated survival time is more than 3 months.
4. At least one assessable tumor lesion (solid tumors according to RECIST 1.1, lymphoma according to Lugano 2014);
5. ECOG physical strength score 0-1;
6. Enough organ function:

   Blood routine (no blood transfusion or colony stimulating factor (G-CSF) treatment within 14 days):ANC≥1.5×109 / L, PLT≥75×109 / L, Hb≥80g/L;Liver function: TBIL≤1.5×ULN, ALT≤2.5×ULN, AST≤2.5×ULN (ALT=5×ULN for liver metastasis patients, AST≤5×ULN);Renal function: Cr ≤ 1.5 × ULN, and creatinine clearance > 50 ml (according to Croft - Gault formula) Coagulation function: activated partial thromboplastin time (APTT) ≤ 1.5 times ULN, prothrombin time (PT) ≤ 1.5 times ULN, international normalized ratio (INR) ≤ 1.5 times ULN;
7. Eligible patients (male and female) with fertility must agree to use reliable methods of contraception (hormone or barrier or abstinence) during the trial period and at least 6 months after the last dose; female patients of childbearing age are selected before the election. The blood or urine pregnancy test within the day must be negative;
8. Prior to the trial, the subject shall have informed consent to the study and voluntarily sign a written form of informed consent;

Exclusion Criteria:

1. Received radiotherapy, chemotherapy, targeted therapy, endocrine therapy or immunotherapy within 4 weeks before the first administration, or other unlisted clinical trial drug therapy (mitomycin and nitrosourea are at least 6 weeks from the last administration, oral fluorouracil drugs such as tegiol and capecitabine are at least 2 weeks from the last administration, and small molecule targeted drugs are at the last administration). At least 2 weeks, or at least 5 half-lives, whichever is longer；
2. Major organ surgery (excluding puncture biopsy) or significant trauma occurred within 4 weeks before the first administration.
3. Adverse reactions of antineoplastic therapy in the past have not been restored to CTCAE grade 5.0≤1 (except for hair loss and other adverse reactions that the investigator judges have no safety risk).
4. Brain metastasis, spinal cord compression, cancerous meningitis with clinical symptoms, or other evidence that the metastasis of brain and spinal cord has not yet been controlled, are not suitable for the group judged by the researchers; patients with suspected clinical symptoms of brain or pia mater diseases need to be excluded by CT/MRI examination;
5. Those who have previously received treatment with PD-1 or PD-L1 inhibitors;
6. In the past, immune-related adverse events (> grade 3) have occurred in immunotherapy (irAE, see Appendix 5)；
7. Patients with active or recurrent autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.)；
8. Current or previous patients with interstitial lung disease;
9. Uncontrolled active infections;
10. History of immunodeficiency, including positive HIV antibody test；
11. Patients with active hepatitis B (HBV titer higher than detection limit) ; hepatitis C virus infection;
12. Those with a history of serious cardiovascular disease;
13. Patients with other serious systemic disease history who are judged to be unsuitable for clinical trials;
14. Alcohol or drug dependence is known;
15. Mental disorder or poor compliance;
16. Pregnant or lactating women;
17. Acceptance of live attenuated vaccine within 4 weeks before the first administration or during the study period is planned.
18. Researchers believe that there are any abnormal clinical or laboratory examinations or other reasons in the subjects and that they are not suitable for this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-04-27 (Actual); Primary Completion 2021-11-26 (Estimated); Study Completion 2022-04-26 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicity (DLT) | At the end of Cycle 1 (28 days).
  An DLT is defined as a ≥Grade 3 drug-related adverse event occurring within the first cycle (28 days) of dosing (excluding tumor flare causing local pain at sites of known or suspected tumor, localized rash, or a transient ≤Grade 3 infusion reaction) using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE).
Maximum tolerable dose (MTD) | At the end of Cycle 1 (28 days).
  MTD refers to the highest dose which can satisfy the first cycle of the same dose group and the proportion of DLT occurring is less than 1/3 in the incremental dose stage. The dose of MTD required confirmation by 6 subjects.

SECONDARY OUTCOMES:
Pharmacokinetic parameters: Observed Maximum Serum Concentration (Cmax) of LDP After Infusion | Up to 22 Days
  Pharmacokinetic parameters Cmax for LDP
Pharmacokinetic Parameters: Area Under the Serum Concentration-time Curve From Time Zero to the Last Sampling Time (AUC0-t) After Infusion AUC(0-t) for LDP | Up to 22 Days
  AUC(0-t) for LDP
Pharmacokinetic parameters: Area Under the Serum Concentration-time Curve From Time Zero to Infinity (AUC0-00) After Infusion Pharmacokinetic parameters: AUC(0-00) for LDP | Up to 22 Days
  Pharmacokinetic parameters: AUC(0-00) for LDP
Pharmacokinetic parameters: Apparent Terminal Half-life (t1/2) of LDP After Infusion | Up to 22 Days
  Pharmacokinetic parameters T1/2 for LDP
Immunogenicity indicators: Number of participants with positive anti-drug antibodies (ADA) | Up to 176 Days
  Immunogenicity indicators: Number of participants with positive anti-drug
Immunogenicity indicators: Number of participants with positive neutralizing antibodies | Up to 176 Days
  Immunogenicity indicators: Number of participants with positive neutralizing antibodies
Objective response rate (ORR) | From first dose of LDP through 21 days after last dose of LDP up to 2 years.
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.
Progression-free survival (PFS) | From first dose of LDP through 21 days after last dose of LDP up to 2 years.
  Progression-free survival is defined as the time from the start of treatment with LDP until the first documentation of disease progression or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Li Jin, doctor, Study Chair — Shanghai East Hospital
Locations (1):
- Dragonboat Biopharmaceutical,Co.,Ltd, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No